CLINICAL TRIAL: NCT02422602
Title: Better Adherence With New Oral Anticoagulant in Atrial Fibrillation : Effectiveness of a Personalized Education Program
Acronym: MONACO
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Montpellier (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 9120
Record Dates: First submitted 2015-04-13; First posted 2015-04-21 (Estimated); Last update posted 2021-07-26 (Actual); Status verified 2020-04

CONDITIONS: Non-valvular Atrial Fibrillation
Keywords: Patients; treated by Rivaroxaban
MeSH Terms: interventions — Rivaroxaban

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (2):
- Taking conventional charge (Active Comparator): No further information is given to the patient during the first and only contact with the nurse of the coordinator center. A time will be dedicated by the IDE to answer questions of the patient.
  Interventions: Drug: Xarelto
- Personalized information intervention (Experimental): The intervention of personalized information will be made as appropriate to the patient's needs and will include: Personalized telephone information carried by a nurse trained in therapeutic education. A time will be dedicated by the IDE to answer questions of the patient. The delivery of paper documents, a list of recommended websites and phone remote monitoring will be performed by the nurse at J30 and J45 to check understanding of the information provided, the actual reading of the paper documents, or effective consultation of websites. A time will be dedicated by the IDE to answer questions at the remote monitoring of the patient to J30 and J45.
  Interventions: Other: Experimental: Personalized information intervention

INTERVENTIONS:
Drug: Xarelto — Taking conventional charge
  Arms: Taking conventional charge
Other: Experimental: Personalized information intervention
  Arms: Personalized information intervention

SUMMARY:
This study is multicentric, single-blind, and interventional with a randomization into two parallel arm, between a standard of care information and an additional information of the patient, with a 12 month follow up.

The aim of this study is to evaluate the effectiveness of a personalized information program versus information provided from standard of care in patients taking Xarelto for Stroke Prevention in Atrial Fibrillation.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated with rivaroxaban chronically, (atrial fibrillation non-valvular under current AMM) for less than one year whatever anti vitamin K treatment history
* Affiliate or beneficiary of a social security system.
* Patient who formulated its "does not oppose" to participate in this research
* Age higher than or equal to 18 years

Exclusion Criteria:

* Opposition to participation
* Patient don't understand french language
* Patient does not have responsibility for the management of treatment (treatment administered by a nurse at home, or by caregivers)
* Tutorship or curatoship
* Law-protected patient
* Pregnant women or breast-feeding

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 196 (Actual)
Dates: Start 2013-11-26 (Actual); Primary Completion 2015-05-06 (Actual); Study Completion 2016-05-06 (Actual)

PRIMARY OUTCOMES:
The occurence of serious adverse event | 12 months
  The occurence of serious adverse event

SECONDARY OUTCOMES:
The number ok hospitalization | 12 months
  The number ok hospitalization

CONTACTS AND LOCATIONS:
Locations (1):
- Heart and vascular diseases service, Montpellier, France